CLINICAL TRIAL: NCT00235352
Title: A Placebo-Controlled Trial of CX516 (Ampakine) Added to Clozapine, Olanzapine or Risperidone in Patients With Schizophrenia
Brief Title: Trial of Ampakine Added to Clozapine, Olanzapine or Risperidone in Patients With Schizophrenia
Acronym: CX516
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: North Suffolk Mental Health Association (Other)
Collaborators: RespireRx (Industry)
Responsible Party: Donald Goff, MD, North Suffolk Mental Health Association
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR43 MH59450
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-02

CONDITIONS: Schizophrenia
Keywords: Schizphrenia; Cognition; Negative Symptoms
MeSH Terms: conditions — Schizophrenia | interventions — 1-(quinoxalin-6-ylcarbonyl)piperidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: CX516 (Ampakine)

SUMMARY:
The purpose of this study is to evaluate the effects of a four-week trial of CX516 900mg tid compared to placebo upon verbal memory, attention and negative symptoms. The AMPA receptor positive modulator, CX516, will be added to a stable dose of clozapine, olanzapine or risperidone in inpatients and outpatients with schizophrenia. The trial is intended to extend and replicate results from our previous placebo-controlled pilot trial of CX516 added to clozapine in which the investigators found improvement in memory and attention (moderate-to-large between group effect sizes) and did not observe serious side effects. Because the investigators' pilot trial also detected at two-week follow-up persistence of cognitive benefits and emergence of a large therapeutic effect upon negative symptoms, this trial will also repeat clinical and cognitive assessments at follow-up, four weeks after completion of the study medication to evaluate persistence and/or strengthening of effects.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Schizophrenia, any subtype
2. Ages 18-65 years
3. Capable of providing informed consent
4. Stable dose of clozapine, olanzapine or risperidone for at least 6 months

Exclusion Criteria:

1. Serious medical or neurological illness (unstable cardiac disease, seizure disorder, malignancy, liver or renal impairment, etc.)
2. Current substance abuse
3. Pregnancy, nursing, or unwilling to use appropriate birth control measures during participation if female and fertile
4. Unable to complete neuropsychological tests
5. History of serious blood dyscrasia requiring discontinuation of clozapine
6. Serious suicidal or homicidal risk within the past six months

Ages: 18 Years to 65 Years
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2002-02; Primary Completion 2005-04 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
1. Evaluate the effects of a four-week trial of CX516 900 mg tid compared to placebo upon verbal memory and attention (DCPT, CVLT, Letter-number sequencing) assessed as part of a standard cognitive battery.
2. Evaluate the effects of CX516 compared to placebo on negative symptoms measured by the SANS total score.
3. Evaluate tolerability and adverse effects measured by the AIMS and SAFTEE Scales.
4. Evaluate persistence and/or strengthening of effects 4 weeks after completion of the 4-week trial.

CONTACTS AND LOCATIONS:
Overall Officials: Donald C Goff, MD, Principal Investigator — North Suffolk Mental Health Association
Locations (1):
- Freedom Trail Clinic, Boston, Massachusetts, United States

REFERENCES:
- [Result] Goff DC, Lamberti JS, Leon AC, Green MF, Miller AL, Patel J, Manschreck T, Freudenreich O, Johnson SA. A placebo-controlled add-on trial of the Ampakine, CX516, for cognitive deficits in schizophrenia. Neuropsychopharmacology. 2008 Feb;33(3):465-72. doi: 10.1038/sj.npp.1301444. Epub 2007 May 9. PMID 17487227